CLINICAL TRIAL: NCT00046332
Title: A Phase II, Randomized, Placebo-controlled Study to Compare Antiviral Effect, Safety, Tolerability and Pharmacokinetics of Four Oral Doses of S-1360 Versus Placebo Over 10 Days in ART-naive HIV-1 Infected Adults.
Brief Title: A Study Comparing 4 Doses Of GW810781 Versus Placebo In HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Shionogi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITG20001
Record Dates: First submitted 2002-09-26; First posted 2002-09-30 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: Integrase inhibitors; Monotherapy; HIV-1 infection
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: GW810781

SUMMARY:
This study will evaluate the drop in viral load over 10 days of treatment with S-1360 versus placebo in HIV-infected patients who have not previously taken anti-HIV medications.

ELIGIBILITY:
Inclusion Criteria:

* No prior HIV medications.
* HIV infection with viral load >400-50,000 copies/mL.
* CD4 cell count >50 cells/mm.

Exclusion Criteria:

* Patients requiring medications that cannot be interrupted for the duration of the study.
* Abnormal ECG or other chronic health conditions as noted on screening physical exam.
* Previous participation in an experimental drug trial(s) within 30 days of the screening visit for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-06; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Plasma HIV-1 RNA change from baseline by Day 11.

SECONDARY OUTCOMES:
HIV-1 RNA slope over 11 days; proportion of subjects with treatment-limiting adverse events; change from baseline in CD4+ cell count at Day 11; plasma pharmacokinetics by dose; emergence of viral resistance.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD,MPH, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Clinical Trials Call Center, Phoenix, Arizona
  - GSK Clinical Trials Call Center, Los Angeles, California
  - GSK Clinical Trials Call Center, San Diego, California
  - GSK Clinical Trials Call Center, San Francisco, California
  - GSK Clinical Trials Call Center, West Hollywood, California
  - GSK Clinical Trials Call Center, Denver, Colorado
  - GSK Clinical Trials Call Center, Washington D.C., District of Columbia
  - GSK Clinical Trials Call Center, Altamonte Springs, Florida
  - GSK Clinical Trials Call Center, Fort Lauderdale, Florida
  - GSK Clinical Trials Call Center, Miami, Florida
  - GSK Clinical Trials Call Center, Tampa, Florida
  - GSK Clinical Trials Call Center, Atlanta, Georgia
  - GSK Clinical Trials Call Center, Indianapolis, Indiana
  - GSK Clinical Trials Call Center, Minneapolis, Minnesota
  - GSK Clinical Trials Call Center, New York, New York
  - GSK Clinical Trials Call Center, The Bronx, New York
  - GSK Clinical Trials Call Center, Chapel Hill, North Carolina
  - GSK Clinical Trials Call Center, Charlotte, North Carolina
  - GSK Clinical Trials Call Center, Durham, North Carolina
  - GSK Clinical Trials Call Center, Dallas, Texas
  - GSK Clinical Trials Call Center, Houston, Texas